CLINICAL TRIAL: NCT03942939
Title: Is TKA With Short Tourniquet Time Superior to TKA With Tourniquet Use in Primary Robotic Assisted TKA? A Prospective, Randomized Study.
Brief Title: Tourniquet vs. Short Time Tourniquet in Primary Robotic Assisted TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Arthur Malkani, Professor, Adult Reconstruction, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19.0365
Record Dates: First submitted 2019-05-03; First posted 2019-05-08 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Knee Arthropathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - TKA with short tourniquet time (Experimental): 50 arms: subjects will receive a tourniquet with a short tourniquet time during TKA surgery. Short tourniquet time is defined in this study as the release of the tourniquet after the initial exposure, resulting in a total tourniquet time of only 10-15 minutes.
  Interventions: Other: Primary Robotic-Assisted Total Knee Arthroplasty with a short tourniquet time
- B - TKA with tourniquet (Active Comparator): 50 arms: subjects will receive a tourniquet during TKA surgery.
  Interventions: Other: Primary Robotic-Assisted Total Knee Arthroplasty with the use of a tourniquet

INTERVENTIONS:
Other: Primary Robotic-Assisted Total Knee Arthroplasty with a short tourniquet time — Primary Robotic-Assisted Total Knee Arthroplasty with a short tourniquet time. Short tourniquet time is defined in this study as the release of the tourniquet after the initial exposure, resulting in a total tourniquet time of only 10-15 minutes.
  Arms: A - TKA with short tourniquet time
Other: Primary Robotic-Assisted Total Knee Arthroplasty with the use of a tourniquet — Primary Robotic-Assisted Total Knee Arthroplasty with the use of a tourniquet
  Arms: B - TKA with tourniquet

SUMMARY:
The goal of this prospective, randomized study is to compare the outcomes of patients undergoing Robotic Arm-Assisted TKA (RA-TKA) with the intraoperative use of a tourniquet to those undergoing RA-TKA with a short tourniquet time.

DETAILED DESCRIPTION:
The goal of this prospective, randomized study is to compare the outcomes of patients undergoing Robotic Arm-Assisted TKA (RA-TKA) with the intraoperative use of a tourniquet to those undergoing RA-TKA with a short tourniquet time. The primary objectives will be to compare the total duration of hospital stay, quadriceps function, and the amount of postoperative narcotics utilized and VAS pain levels. The secondary objective will be to compare variables of patient functionality at five postoperative intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over the age of 21
2. Patient is scheduled to undergo a unilateral, cementless primary RA-TKA, secondary to osteoarthritis
3. Surgical approach is subvastus approach
4. Patient's BMI (body mass index) is less than 40 at time of surgery.
5. Patient agrees to participate as a study subject and signs the Informed Consent and Research Authorization documents
6. Patient is able to read and speak English

Exclusion Criteria:

1. Patient is under the age of 21
2. Patient's primary diagnosis is not osteoarthritis (e.g. post-traumatic arthritis)
3. Patient is scheduled to undergo a bilateral TKA surgery
4. Patient BMI is > 40
5. Patient is unable to read and speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery)
  Knee Society Score. The score is on a scale from 0-100. A higher value represents a better outcome.
Knee Society Score | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Knee Society Score. The score is on a scale from 0-100. A higher value represents a better outcome.
Knee Society Score | outcome measure will be taken 1 year (± 2 months) postoperatively
  Knee Society Score. The score is on a scale from 0-100. A higher value represents a better outcome.
WOMAC Score | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery)
  WOMAC score. The score is on a scale from 0-100. In contrast to the Knee Society Score, on the WOMAC a lower value represents a better outcome.
WOMAC Score | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  WOMAC score. The score is on a scale from 0-100. In contrast to the Knee Society Score, on the WOMAC a lower value represents a better outcome.
WOMAC Score | outcome measure will be taken 1 year (± 2 months) postoperatively
  WOMAC score. The score is on a scale from 0-100. In contrast to the Knee Society Score, on the WOMAC a lower value represents a better outcome.
Active range-of-motion (ROM) | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery)
  Active ROM (range-of-motion) as measured by a goniometer (range of 0-135 degrees)
Active range-of-motion (ROM) | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Active ROM (range-of-motion) as measured by a goniometer (range of 0-135 degrees)
Active range-of-motion (ROM) | outcome measure will be taken 1 year (± 2 months) postoperatively
  Active ROM (range-of-motion) as measured by a goniometer (range of 0-135 degrees)
Amount of narcotic medication utilized | outcome measure will be taken 24 hours postoperatively
  Amount of narcotic medication utilized (daily dosage measured as a Milligram Morphine Equivalent (MME) value).
Amount of narcotic medication utilized | outcome measure will be taken 48 hours postoperatively
  Amount of narcotic medication utilized (daily dosage measured as a Milligram Morphine Equivalent (MME) value).
Amount of narcotic medication utilized | outcome measure will be taken 72 hours postoperatively
  Amount of narcotic medication utilized (daily dosage measured as a Milligram Morphine Equivalent (MME) value).
Amount of narcotic medication utilized | outcome measure will be taken 2 weeks (± 4 days) postoperatively
  Amount of narcotic medication utilized (daily dosage measured as a Milligram Morphine Equivalent (MME) value).
Amount of narcotic medication utilized | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Amount of narcotic medication utilized (daily dosage measured as a Milligram Morphine Equivalent (MME) value).
Visual Analog Scale | outcome measure will be taken 24 hours postoperatively
  The Visual Analog Scale measures the patient's level of knee pain on a scale of zero to ten via what the patient expresses verbally. The Visual Analog Scale (VAS) represents the degree of pain that the patient is experiencing at the time the measure is taken. Zero represents "pain-free". A 10 would represent pain so excruciating as to warrant emergency medical assistance, or as it is described to the patient, "the worst pain imaginable". Obviously, the lower the number, the better the outcome. There is no subscale.
Visual Analog Scale | outcome measure will be taken 48 hours postoperatively
  The Visual Analog Scale measures the patient's level of knee pain on a scale of zero to ten via what the patient expresses verbally. The Visual Analog Scale (VAS) represents the degree of pain that the patient is experiencing at the time the measure is taken. Zero represents "pain-free". A 10 would represent pain so excruciating as to warrant emergency medical assistance, or as it is described to the patient, "the worst pain imaginable". Obviously, the lower the number, the better the outcome. There is no subscale.
Visual Analog Scale | outcome measure will be taken 72 hours postoperatively
  The Visual Analog Scale measures the patient's level of knee pain on a scale of zero to ten via what the patient expresses verbally. The Visual Analog Scale (VAS) represents the degree of pain that the patient is experiencing at the time the measure is taken. Zero represents "pain-free". A 10 would represent pain so excruciating as to warrant emergency medical assistance, or as it is described to the patient, "the worst pain imaginable". Obviously, the lower the number, the better the outcome. There is no subscale.
Visual Analog Scale | outcome measure will be taken 2 weeks (± 4 days) postoperatively
  The Visual Analog Scale measures the patient's level of knee pain on a scale of zero to ten via what the patient expresses verbally. The Visual Analog Scale (VAS) represents the degree of pain that the patient is experiencing at the time the measure is taken. Zero represents "pain-free". A 10 would represent pain so excruciating as to warrant emergency medical assistance, or as it is described to the patient, "the worst pain imaginable". Obviously, the lower the number, the better the outcome. There is no subscale.
Visual Analog Scale | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  The Visual Analog Scale measures the patient's level of knee pain on a scale of zero to ten via what the patient expresses verbally. The Visual Analog Scale (VAS) represents the degree of pain that the patient is experiencing at the time the measure is taken. Zero represents "pain-free". A 10 would represent pain so excruciating as to warrant emergency medical assistance, or as it is described to the patient, "the worst pain imaginable". Obviously, the lower the number, the better the outcome. There is no subscale.
Distance that patient is able to walk | outcome measure will be taken 24 hours postoperatively
  Distance that patient is able to walk, as measured in feet
Distance that patient is able to walk | outcome measure will be taken 48 hours postoperatively
  Distance that patient is able to walk, as measured in feet
Distance that patient is able to walk | outcome measure will be taken 72 hours postoperatively
  Distance that patient is able to walk, as measured in feet
Distance that patient is able to walk | outcome measure will be taken 2 weeks (± 4 days) postoperatively
  Distance that patient is able to walk, as measured in feet
Distance that patient is able to walk | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Distance that patient is able to walk, as measured in feet
Ability to rise from a chair independently | outcome measure will be taken 24 hours postoperatively
  Ability to rise from a chair independently (Yes/No)
Ability to rise from a chair independently | outcome measure will be taken 48 hours postoperatively
  Ability to rise from a chair independently (Yes/No)
Ability to rise from a chair independently | outcome measure will be taken 72 hours postoperatively
  Ability to rise from a chair independently (Yes/No)
Ability to rise from a chair independently | outcome measure will be taken 2 weeks (± 4 days) postoperatively
  Ability to rise from a chair independently (Yes/No)
Ability to rise from a chair independently | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Ability to rise from a chair independently (Yes/No)
Use of an ambulatory assistive device | outcome measure will be taken 24 hours postoperatively
  Use of an ambulatory assistive device (Yes/No)
Use of an ambulatory assistive device | outcome measure will be taken 48 hours postoperatively
  Use of an ambulatory assistive device (Yes/No)
Use of an ambulatory assistive device | outcome measure will be taken 72 hours postoperatively
  Use of an ambulatory assistive device (Yes/No)
Use of an ambulatory assistive device | outcome measure will be taken 2 weeks (± 4 days) postoperatively
  Use of an ambulatory assistive device (Yes/No)
Use of an ambulatory assistive device | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Use of an ambulatory assistive device (Yes/No)
Return to driving | outcome measure will be taken 2 weeks (± 4 days) postoperatively
  Return to driving (Yes/No)
Return to driving | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Return to driving (Yes/No)
Level of Patient Satisfaction: 5-point Likert scale | outcome measure will be taken at 6 weeks (± 2 weeks) postoperatively.
  Level of Patient Satisfaction as measured using a 5-point Likert scale
Level of Patient Satisfaction: 5-point Likert scale | outcome measure will be taken 1 year (± 2 months) postoperatively
  Level of Patient Satisfaction as measured using a 5-point Likert scale
Quadriceps Function | outcome measure will be taken at 2 weeks (± 4 days)
  Quadriceps Function as measured in peak force in kilograms by a Hand-held dynamometer (model 01163; Lafayette Instrument Company, Lafayette, Ind., USA)
Quadriceps Function | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Quadriceps Function as measured in peak force in kilograms by a Hand-held dynamometer (model 01163; Lafayette Instrument Company, Lafayette, Ind., USA)
Quadriceps Function | outcome measure will be taken 1 year (± 2 months) postoperatively
  Quadriceps Function as measured in peak force in kilograms by a Hand-held dynamometer (model 01163; Lafayette Instrument Company, Lafayette, Ind., USA)
total length of hospital stay | outcome measure will be taken at 2 weeks postoperatively
  total length of hospital stay as defined by number of days from date of surgery to date of discharge
Dates of postoperative exams | outcome measure will be taken at 2 weeks (± 4 days) postoperatively
  Dates of postoperative exams as defined by dates that subject returns to the P.I.'s office for postoperative exam
Dates of postoperative exams | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Dates of postoperative exams as defined by dates that subject returns to the P.I.'s office for postoperative exam
Dates of postoperative exams | outcome measure will be taken 1 year (± 2 months) postoperatively
  Dates of postoperative exams as defined by dates that subject returns to the P.I.'s office for postoperative exam
Incidence of postop transfusion | outcome measure will be taken at 2 weeks postoperatively
  Incidence of postop transfusion as defined by one or more transfusions of blood to the subject postoperatively
Change in creatinine level (CKMB) | outcome measures will be taken preoperatively (4-6 weeks prior to date of surgery) and on postoperative day number two.
  Change in CKMB (creatinine level) as defined by the CKMB values recorded in the participant's lab report
Change in hemoglobin level (HgB) | outcome measures will be taken preoperatively (4-6 weeks prior to date of surgery) and on postoperative day number two.
  Change in HgB as defined by the HgB values recorded in the participant's lab report
Operative Time | outcome measure will be taken at 2 weeks postoperatively
  Total Operative Time as defined in minutes
Estimated Blood Loss (EBL) | outcome measure will be taken at 2 weeks postoperatively
  Estimated Blood Loss as defined by the amount of intraoperative blood loss measured in cubic centimeters (cc).

SECONDARY OUTCOMES:
Number of Participants with postoperative complications | outcome measure will be taken at 1 year (± 2 months) postoperatively
  Number of Participants with postoperative complications. A postoperative complication is defined as any diagnosis or condition that necessitates a re-operation on the surgical knee

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L Malkani, MD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No